CLINICAL TRIAL: NCT04442750
Title: Comparison of the Analgesic Efficacy of Three Different Concentrations of Bupivacaine in Ultrasound Guided Erector Spinae Plane Block in Hip Surgeries: Randomized Control Trial
Brief Title: Different Concentrations of Bupivacaine in Erector Spinae Plane Block in Hip Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N-29-2020
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (0.5%) group (Experimental): patients will receive a single shot erector spinae block with 30 ml 0.5% bupivacaine followed by general anesthesia
  Interventions: Procedure: Erector spinae plane block Technique; Procedure: General anesthesia; Drug: Bupivacaine 0.5%
- B (0.375%) group (Experimental): patients will receive a single shot erector spinae block with 30 ml 0.375% bupivacaine followed by general anesthesia
  Interventions: Procedure: Erector spinae plane block Technique; Procedure: General anesthesia; Drug: Bupivacaine 0.375%
- C (0.25%) group (Experimental): patients will receive a single shot erector spinae block with 30 ml 0.25% bupivacaine followed by general anesthesia
  Interventions: Procedure: Erector spinae plane block Technique; Procedure: General anesthesia; Drug: Bupivacaine 0.25%

INTERVENTIONS:
Procedure: Erector spinae plane block Technique — The patient will be placed in Lateral Decubitus with a surgical side upwards. A curvilinear array ultrasound probe will be placed in a transverse orientation at L4 level to identify the tip of the L4 transverse process. The tip of the transverse process will be centered on the ultrasound screen and the probe will be then rotated into a longitudinal orientation 2-3 cm lateral to vertebral column. The lumbar skin region will be sterilized, local infiltration of the skin and subcutaneous tissue will be applied by 2-3ml of lidocaine 2%. Then, using ultrasound guidance, A 38-mm 22-gauge (22-G, 50-mm 'Stimuplex A'; BBraun, Melsung, Germany) regional block needle will be advanced in plane to the ultrasound beam in a cranial-to-caudal direction until contact will made with the L4 transverse process. Local anesthetic solution will be injected and its type will be selected according to the studied group and patients were placed in a supine position and general anesthesia will be started.
Procedure: General anesthesia — Induction of general anaesthesia will be performed using a regimen of IV 2 μg/kg fentanyl and propofol IV 2 mg /kg. Tracheal intubation will be facilitated using 0.5 mg/kg IV of rocuronium.
  Anaesthesia will be maintained with inhaled sevoflurane 1-1.5% in oxygen enriched air (FiO2=0.5). Maintenance doses of rocuronium o.1 m\kg will be provided every 30 minutes.
  Rescue analgesia of fentanyl 1 μg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels.
  At the end of surgery, residual neuromuscular blockade will be reversed using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg), and will extubation be performed after complete recovery of the airway reflexes.
Drug: Bupivacaine 0.5% — The patient will receive 30ml bupivacain 0.5% in erector spinae block
  Arms: A (0.5%) group
Drug: Bupivacaine 0.375% — The patient will receive 30ml bupivacain 0.375% in erector spinae block
  Arms: B (0.375%) group
Drug: Bupivacaine 0.25% — The patient will receive 30ml bupivacain 0.25% in erector spinae block
  Arms: C (0.25%) group

SUMMARY:
The prevalence of hip replacement surgery is increasing nowadays. Patients are usually older age and suffer from comorbidities may be an anesthetic and analgesic challenge. Erector spinae plane block (ESPB) is a newly described technique that is has been demonstrated in previous studies for chronic and acute pain treatment. The exact volume and concentration of local anesthetic (LA) to be used in ESPB is not well established.

DETAILED DESCRIPTION:
Aim of the work is to compare the analgesic effects of three different concentrations of the same volume of local anesthetics; 30 ml of 0.50% vs 0.375% vs 0.25% bupivacaine in patients undergoing hip surgeries.

Prospective randomized double blinded study that will be conducted in at Kasr El-Ainy hospital orthopedic surgical theater.

patients, undergoing hip surgeries will be randomly allocated into three equal groups, each (n=44), using computerized generated random tables

1. Group F: 44 patients will receive single shot erector spinae block at the level of L4 with 30 ml 0.50% bupivacaine.
2. Group M: 44 patients will receive single shot erector spinae block at the level of L4 with 30 ml 0.375% bupivacaine.
3. Group H: 44 patients will receive single shot of erector spinae block at the level of L4with 30ml 0.25% bupivacaine .

ELIGIBILITY:
Inclusion Criteria:

* Both genders (Males and females).
* Type of surgery; unilateral elective hip surgeries
* Physical status ASA I, II.
* Age ≥ 18 and ≤ 65 Years.
* Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.

Exclusion Criteria:

* Patients with known sensitivity or contraindication to drug used in the study (local anesthetics, opioids).
* History of psychological disorders and/or chronic pain.
* Contraindication to regional anesthesia e.g. local sepsis, pre- existing peripheral neuropathies and coagulopathy.
* Infection of the skin at the site of needle puncture area.
* Patient refusal.
* Severe respiratory or cardiac disorders.
* Advanced liver or kidney disease.
* Pregnancy.
* Patient with surgery duration more than two hours.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-10-20 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
The total 24 hours amount of morphine consumption | 24 hours postoperative
  The total amount of morphine consumption in the first 24 hours postoperatively

SECONDARY OUTCOMES:
Total amount of intraoperative fentanyl | 2 hours intraoperatively
Numeric Pain Rating Scale | 24 hours postoperative
  Numeric Pain Rating Scale, both at rest and during movement: 30 minutes,2, 4,6, 8, 12, 16, 20 and 24 hours postoperatively. The Numeric Rating Scale (NRS) is the simplest and most commonly used numeric scale in which the patient rates the pain from 0 (no pain) to 10 (worst pain).
Time for first rescue analgesia | 24 hours
Block related complications | 24 hours postoperative
  • Block related complications such as local anesthetic toxicity, hematoma formation and lower limb weakness.

CONTACTS AND LOCATIONS:
Overall Officials: Bassant abdelhamid, M.D., Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Selvi O, Senturk O, Ermis MN, Cubuk R, Ozer Z. Clinical experiences of ultrasound-guided lumbar erector spinae plane block for hip joint and proximal femur surgeries. J Clin Anesth. 2018 Jun;47:5-6. doi: 10.1016/j.jclinane.2018.02.014. Epub 2018 Mar 6. No abstract available. PMID 29522966
- [Background] Tulgar S, Kose HC, Selvi O, Senturk O, Thomas DT, Ermis MN, Ozer Z. Comparison of Ultrasound-Guided Lumbar Erector Spinae Plane Block and Transmuscular Quadratus Lumborum Block for Postoperative Analgesia in Hip and Proximal Femur Surgery: A Prospective Randomized Feasibility Study. Anesth Essays Res. 2018 Oct-Dec;12(4):825-831. doi: 10.4103/aer.AER_142_18. PMID 30662115
- [Background] Kashani HH, Grocott HP. Clarity needed as to the optimal dose and volume of local anesthetic for erector spinae plane blockade for posterior rib fractures. Am J Emerg Med. 2018 Jun;36(6):1102-1103. doi: 10.1016/j.ajem.2018.03.032. Epub 2018 Mar 15. No abstract available. PMID 29576256